CLINICAL TRIAL: NCT03628508
Title: External Tibia Torsion and Passive Muscle Stiffness of Quadriceps as Two Important Contributors of Joint Loading During Walking in People With Knee Osteoarthritis
Brief Title: Muscle Property, Alignment and Joint Loading in People With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20170406003
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee
Keywords: muscle tension; alignment; knee osteoarthritis; loading
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Six-week exercise including stretching, strengthening, endurance and gait modification
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Comprehensive exercise program including strengthening, stretching, gait modification etc.

SUMMARY:
Knee osteoarthritis (KOA) is a common chronic painful musculoskeletal condition among older adults. It poses great challenge to the health care system due to its inability to be cured. Understanding factors associated with disease progression in KOA should assist the development of novel prevention/rehabilitation strategies. This study investigate factors including muscle properties, lower limb alignment and joint loading in patients with knee osteoarthritis before and after a six-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-80
2. having radiographic tibiofemoral joint OA in the medial compartment defined as Kellgren and Lawrence grade = 2 to 3
3. having medial knee pain on most days of the month
4. having a minimum average pain score of 2 on an 11-point numerical rating scale in the past week while walking

Exclusion Criteria:

1. having lateral tibiofemoral compartment osteophytes greater than the medial side.
2. having undergone intra-articular corticosteroid injection or knee surgery to either knee within the past 3 months
3. having a systemic arthritic condition (e.g., rheumatoid arthritis)
4. having a knee joint replacement or high tibial osteotomy in the past
5. having any other muscular, joint or neurological condition influencing lower limb function
6. unable to walk unaided
7. having low back, hip, ankle or foot pain > 3 on numerical rating scale
8. having a body mass index (BMI) >36 kg/ m2

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siu Ngor Fu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 40
Completed | 39
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 40

OUTCOME MEASURES:

1. Primary Outcome: Change of External Knee Adduction Moment as Assessed by Visual Motion Analysis System
Description: External knee moment in the frontal plane during early stance phase of walking
Time Frame: At baseline and one week after intervention
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Exercise
Number analyzed (Participants) | 40
Nm/kg | 0.50 (0.13)

2. Secondary Outcome: Change of Pain Severity Score as Assessed by Knee Injury and Osteoarthritis Outcome Score
Description: Pain intensity measured by the pain subscale of Knee injury and Osteoarthritis Outcome Score (KOOS). The minimum value is 0 and maximum value is 100. The higher scores mean a better outcome.
Time Frame: At baseline and one week after intervention
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exercise
Number analyzed (Participants) | 39
Score on a scale | 70 (14)

3. Secondary Outcome: Tibial Torsion as Assessed by X-ray Imaging
Description: The angle between tibial and femur in the transverse plane
Time Frame: At baseline
Reporting Status: Not Posted

4. Secondary Outcome: Change of Young's Modulus of Quadriceps as Assessed by Ultrasound Elastography
Description: Young's modulus by ultrasound elastography
Time Frame: At baseline and one week after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks since start of exercise program 1 year after finishing the exercise program
Arm/Group | Exercise
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03628508/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03628508/ICF_001.pdf